CLINICAL TRIAL: NCT03593759
Title: Cardiac Sarcoidosis Multi-Center Randomized Controlled Trial
Brief Title: Cardiac Sarcoidosis Randomized Trial
Acronym: CHASM-CS-RCT
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Ottawa Heart Institute Research Corporation (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: UOttawaHI
Record Dates: First submitted 2018-06-27; First posted 2018-07-20 (Actual); Last update posted 2024-12-03 (Actual); Status verified 2024-10

CONDITIONS: Cardiac Sarcoidosis; Sarcoidosis
Keywords: Cardiac Sarcoidosis; Prednisone (or Prednisolone); Methotrexate
MeSH Terms: conditions — Sarcoidosis | interventions — Prednisone; Prednisolone; Methotrexate

STUDY DESIGN:
Intervention Model Description: Prospective, open-label, non-inferiority, randomized controlled with blinded end-point analysis.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Prednisone (or Prednisolone) (Active Comparator): [Dose everywhere except Japan] Prednisone 0.5 mg kg/day for 6 months (max dose 30 mg)
  [Dose in Japan] Prednisone or prednisolone 0.5 mg/kg po (max 30mg) for one month then reduce by 5 mg per month for five months
  Interventions: Drug: Prednisone or Prednisolone
- Methotrexate (Experimental): [Dose everywhere except Japan] Methotrexate 15-20 mg orally, sc, or IM once a week for 6 months + Prednisone 20 mg po daily for one month then 10 mg po daily for one month then 5 mg po daily for one month and then stop. Also Folic Acid OD (exact dose and directions at physicians discretion) for 6 months.
  [Dose in Japan] Methotrexate 5-20mg mg orally, sc, or IM once a week for 6 months+ Prednisone or Prednisolone 20mg OD for 1 month then 10mg OD for 1 month then 5 mg OD one month. Also Folic Acid 2 mg po daily for 6 months.
  Interventions: Drug: Prednisone or Prednisolone; Drug: Methotrexate

INTERVENTIONS:
Drug: Prednisone or Prednisolone — Oral prednisone/prednisolone tablet
Drug: Methotrexate — Oral, subcutaneous, or intramuscular methotrexate
  Arms: Methotrexate

SUMMARY:
Prospective randomized controlled trial comparing low dose Prednisone(or Prednisolone)/Methotrexate combination to standard dose Prednisone(or Prednisolone) in patients diagnosed with acute active clinically manifest cardiac sarcoidosis and not yet treated.

The Investigators hypothesize that low dose Prednisone(or Prednisolone)/Methotrexate combination will be as effective as standard dose Prednisone(or Prednisolone), and result in significantly better quality of life and less toxicity than standard dose Prednisone(or Prednisolone).

DETAILED DESCRIPTION:
Subjects meeting the study inclusion/exclusion criteria will be randomized equally to receive either:

Everywhere but Japan:

1. Prednisone 0.5 mg kg/day for 6-months (MAX dose 30 mg per day) or
2. Methotrexate 15-20 mg po, sc, or IM once a week for 6-months + Folic Acid OD (exact dose and directions at physician) for 6 months + Prednisone 20 mg day for 1 month, then 10 mg OD for 1 month, then 5 mg OD for one month then STOP

In Japan:

1. Prednisone or prednisolone 0.5 mg/kg po (max 30mg) for one month then reduce by 5 mg per month for five months or
2. Methotrexate 5-20mg po, sc or IM once week for 6-months +Folic Acid 2-5 mg OD for 6-months+Prednisone or prednisolone 20mg OD for 1 month then 10mg OD for 1 month then 5 mg OD one month

Methotrexate will be initiated at a dose of 15 mg once a week and increased to 20 mg once a week after 4 weeks if tolerated. In case of Methotrexate-induced side-effects general guidelines will be provided, however specific management will be left to the treating physicians. Folic acid will be taken to help reduce methotrexate side-effects.

Prior to randomization and study treatment all subjects will have the following baseline tests done: baseline safety blood work; FDG-PET scan with myocardial perfusion imaging; ECG; echo; and an optional bone mineral density scan. Cardiac MRI (CMR) is optional but strongly encouraged. Blood will be obtained for biomarker core-lab analysis. Biomarkers to be assayed will include highly sensitive Troponin I. Samples will be stored for future novel biomarker discovery. Quality of LIfe (QOL) questionnaires (KSQ, SAT and SF-36) will be completed prior to treatment start.

After therapy initiation subjects will be seen at 4 weeks, 8 weeks (methotrexate arm only), and 12 weeks, with a final visit at 6 months. Safety bloodwork and assessment for medication side effects, using a medication side-effect questionnaire, will be completed at all visits. At 12 weeks QOL questionnaires will be completed. The primary endpoint will be assessed at 6-months, when FDG-PET with myocardial perfusion imaging, ECG, echo, optional bone mineral density scan, QOL questionnaires, blood for biomarkers and device interrogation will be done. CMR may be repeated. Skin, muscle strength testing and neuropsychiatric assessment will be completed at 6 months as part of the composite glucocorticoid toxicity index.

After the 6 month visit. further management will be at the treating physician's discretion. Details of the physicians planned treatment following the 6-month PET scan will be collected.

Standardized protocols for all aspects of FDG-PET scans (i.e. patient preparation, image acquisition, image processing, transfer to the core lab and analysis at core lab) will be followed.

ELIGIBILITY:
Inclusion Criteria:

(i) Cardiac sarcoidosis presenting with one or more of the following clinical findings:

* advanced conduction system disease (defined as Mobitz II AV block or third degree AV block)
* significant sinus node dysfunction (defined as average HR less than 40bpm when awake and/or sustained atrial arrhythmias)
* non- sustained or sustained ventricular arrhythmia
* left ventricular dysfunction (LVEF < 50%)
* right ventricular dysfunction (RVEF < 40%)

AND

(ii) No alternative explanation for clinical features

AND

(iii) Nuclear Imaging within six-months of enrollment consisting of FDG-PET scan with FDG uptake suggestive of active CS and myocardial perfusion imaging

AND ONE OR BOTH OF FOLLOWING

(iv) Positive biopsy for Sarcoid (either EMB or extra-cardiac)

(v) CT Chest showing features consistent with pulmonary sarcoidosis and/or mediastinal and/or hilar lymphadenopathy

Exclusion Criteria:

1. Current or recent (within two months) non-topical treatment for sarcoidosis
2. Current Oral/IV treatment of duration greater than 5 days
3. Currently taking Methotrexate or Prednisone for another health condition
4. Intolerance or contra-indication to Methotrexate or Prednisone
5. Patient does not meet all of the above listed inclusion criteria
6. Patient is unable or unwilling to provide informed consent
7. Patient is included in another randomized clinical trial
8. Patient has a contraindication to PET imaging or is unlikely to tolerate due to severe claustrophobia
9. Pregnancy (all women of child bearing age and potential will have a negative BHCG test before enrollment)
10. Breastfeeding
11. Women of childbearing age who refuse to use a highly effective and medically acceptable form of contraception throughout the study
12. Patients for whom the investigator believes that the trial is not in the interest of the patient

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 194 (Estimated)
Dates: Start 2019-01-15 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Summed perfusion rest score (SPRS) on FDG-PET scan | 6 months
  Measure of myocardial scarring and fibrosis (blinded core lab analysis)

SECONDARY OUTCOMES:
Mortality | 6 months
  All cause deaths
Cardiovascular hospitalizations | 6 months
  Cardiovascular related only
Medication related adverse events | 6 months
  Using clinical assessment, medication side-effect and adverse event reporting
Modified Cleveland Clinic Glucocorticoid Toxicity Score | 6 months
  Summed score of new/worsening diabetes;new/worsening HTN; osteoporosis; change in height and weight (combined and reported as BMI in kg/m2)
Glucocorticoid Toxicity Index | 6 months
  Composite scoring (improvement; no significant change; worsening) compared to baseline
Patient reported symptoms related to medication | 6 months
  Using medication side-effect questionnaire ( symptom present, yes or no; frequency; intensity)
Medication compliance | 6 months
  % of days where treatment was taken as prescribed
Generic Quality of Life (SF 36) | 6 months
  Measuring general QOL using SF-36 questionnaire
Disease Specific Quality of Life (KSQ and SAT) | 6 months
  Using Kings Sarcoidosis questionnaire and Sarcoidosis Assessment Tool
BMI | 6 months
  Weight and height combined to report BMI in kg/m2, absolute and delta compared to baseline
Blood pressure | 6 months
  Systolic and diastolic, absolute and delta compared to baseline
HbA1C | 6 months
  Absolute and delta compared to baseline
T-score on bone density scan | 6 months
  Absolute and delta compared to baseline
FDG-PET and myocardial perfusion | 6 month scan
  SPRS in mismatched segments; SUVmax, SUVmean and COI; LVEF, RVEF; whole body disease activity
Ventricular arrhythmia burden | 6 months
  Episodes of sustained ventricular arrhythmia or episodes requiring appropriate ICD therapy (shock or anti-tachycardia pacing)
Complete heart block | 6 months
  Percentage of patients who are in CHB
LVEF and RVEF assessed on echocardiogram | 6 months
  Ejection fraction, absolute and delta compared to baseline
Highly sensitive Troponin I levels and BNP levels | 6 months
  Absolute and delta compared to baseline
CMR Endpoints | 6 months
  Volume of delayed enhancement

CONTACTS AND LOCATIONS:
Overall Officials: David H Birnie, MD, Principal Investigator — Ottawa Heart Institute Research Corporation
Locations (30):
- United States (9):
  - Yale-New Haven Hospital, New Haven, Connecticut
  - Tufts Medical Center, Boston, Massachusetts
  - University of Michigan-Michigan Medicine Cardiovascular Center, Ann Arbor, Michigan
  - University of Minnesota, Minneota, Minnesota
  - Montefiore Medical Center, New York, New York
  - The Ohio State University Wexner Medical Center, Columbus, Ohio
  - Allegheny General Hospital, Pittsburgh, Pennsylvania
  - University of Utah, Salt Lake City, Utah
  - Virginia Commonwealth University, Richmond, Virginia
- Canada (11):
  - Libin Cardiovascular Institute of Alberta, Calgary, Alberta
  - St. Paul's Hospital, Vancouver, British Columbia
  - Eastern Health Health Sciences Centre, St. John's, Newfoundland and Labrador
  - QE II Health Sciences Centre, Halifax, Nova Scotia
  - St. Joseph's Healthcare Centre, Hamilton, Ontario
  - London Health Sciences Centre, London, Ontario
  - University of Ottawa Heart Institute, Ottawa, Ontario
  - Montreal Heart Institute, Montreal, Quebec
  - CIUSSS-Hopital du Sacre-Coeur de Montreal, Montreal, Quebec
  - Institut universitaire de cardiologie et de pneumologie de Québec-Université Laval, Québec, Quebec
  - CIUSSS de l'Estrie - CHUS - Hôpital Fleurimont, Sherbrooke, Quebec
- Japan (8):
  - Hokkaido University, Sapporo, Kita 8, Nishi 5, Kita-Ku
  - Chiba University, Chiba
  - University of Fukui, Fukui
  - St. Marrianna University, Kawasaki
  - Nagoya City University, Nagoya
  - National Cerebral and Cardiovascular Center (NCVC), Osaka
  - Sapporo Medical University, Sapporo
  - Nippon Medical School, Tokyo
- United Kingdom (2):
  - King's College Hospital NHS Foundation Trust, London
  - Imperial College Healthcare Trust-NHS-Hammersmith Hospital, London

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Birnie D, Beanlands RSB, Nery P, Aaron SD, Culver DA, DeKemp RA, Gula L, Ha A, Healey JS, Inoue Y, Judson MA, Juneau D, Kusano K, Quinn R, Rivard L, Toma M, Varnava A, Wells G, Wickremasinghe M, Kron J. Cardiac Sarcoidosis multi-center randomized controlled trial (CHASM CS- RCT). Am Heart J. 2020 Feb;220:246-252. doi: 10.1016/j.ahj.2019.10.003. Epub 2019 Oct 20. PMID 31911261